CLINICAL TRIAL: NCT05062460
Title: Adherence to One- Versus Two-hour Postprandial Glucose Monitoring in Gestational Diabetics: A Randomized Trial
Brief Title: Glucose Testing in GDM: Adherence to One- Versus Two-hour Postprandial Glucose Monitoring in Gestational Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-10022829
Record Dates: First submitted 2021-08-19; First posted 2021-09-30 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Blood Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1-hour post-prandial blood glucose monitoring Arm (Other): Arm in which participants are randomized to blood glucose monitoring at 1 hour after eating.
  Interventions: Other: 1 hour Blood glucose monitoring
- 2-hour post-prandial blood glucose monitoring Arm (Other): Arm in which participants are randomized to blood glucose monitoring at 2 hours after eating.
  Interventions: Other: 2 hour blood glucose monitoring

INTERVENTIONS:
Other: 1 hour Blood glucose monitoring — Consented patients who are diagnosed with gestational diabetes will be randomized to 1-hour postprandial blood glucose monitoring.
  Arms: 1-hour post-prandial blood glucose monitoring Arm
Other: 2 hour blood glucose monitoring — Consented patients who are diagnosed with gestational diabetes will be randomized to 2 hour post prandial blood glucose monitoring
  Arms: 2-hour post-prandial blood glucose monitoring Arm

SUMMARY:
The purpose of this study is to evaluate if in patients with gestational diabetes (GDM), adherence to postprandial glucose monitoring differs when performed 1-hour versus 2-hours after eating.

The primary objective of this study is to evaluate difference in rate of adherence (binary outcome defined as <80% or ≥80% of glucose log completed) between gestational diabetics who perform 1-hour versus 2-hour postprandial blood glucose testing.

DETAILED DESCRIPTION:
Consented patients who are diagnosed with gestational diabetes will be randomized to either 1-hour or 2-hour postprandial blood glucose monitoring. A retrospective chart review from July 2020 until study commencement for patients from the same clinic will be used as a historical control group. This study will assess differences in adherence to testing.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients with singleton gestation who are ≥ 18 years of age.
* Diagnosis of GDM after 24 0/7 weeks.
* For diagnosing GDM, a two-step screening algorithm will be performed according to the American College of Obstetrics and Gynecologists.4 Specifically, a 1-hour 50-g glucose-loading test is given first. Plasma glucose levels between 140 and 200 mg/dL will be considered elevated. Confirmatory testing will then be performed using a 3-hour 100-g glucose tolerance test. Diagnosis was made when two of the four values were elevated. Abnormal glucose value thresholds are established via the criteria suggested by Carpenter and Coustan: fasting value ≥ 95 mg/dL, 1-hour ≥ 180 mg/dL, 2-hour ≥ 155 mg/dL, and 3-hour ≥ 140 mg/dL.9 Patients with a blood glucose level greater than 200 mg/dL after 1-hour 50-g glucose-loading test will be diagnosed with GDM without requirement for the 3-hour 100-g glucose tolerance test.

Exclusion Criteria:

* Type 1 pre-gestational diabetes
* Type 2 pre-gestational diabetes
* GDM diagnosed prior to 24 0/7 weeks gestation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Rate of adherence | During the intervention
  Evaluate rate of adherence (binary outcome defined as <80% or ≥80% of glucose log completed) between gestational diabetics who perform 1-hour versus 2-hour postprandial blood glucose testing.

SECONDARY OUTCOMES:
Percentage of postprandial glucose log complete, averaged over the duration of the study period | During the intervention
Percentage of postprandial glucose log complete for each meal (breakfast, lunch, and dinner), averaged over the duration of the study period | During the intervention
Percentage of elevated blood glucose values per week, averaged over the duration of the study period | During the intervention
Number of patients who start insulin or oral hyperglycemic medication therapy prior to delivery. | During the intervention
Gestational age at medication therapy initiation | During the intervention
Timeframe from diagnosis of gestational diabetes to initiation of insulin therapy | During the intervention
Number of subjects with a vaginal delivery | At time of delivery
Number of subjects with an operative delivery | At time of delivery
Number of subjects with a caesarean section delivery | At time of delivery
Number of subjects with a preeclampsia diagnosis | During intervention
Neonatal birthweight | At time of delivery
Number of subjects with shoulder dystocia | At time of delivery
Number of patients with 3rd or 4th degree perineal lacerations | At time of delivery
Number of patients with postpartum hemorrhage. | At time of delivery
Number of stillbirths | At time of delivery
Number of NICU admissions | At time of delivery
Number of patients requiring supplemental oxygen support | At time of delivery
Number of patients with diagnosis of hypoglycemia | At time of delivery
Number of patients with diagnosis of hyperbilirubinemia | At time of delivery
Number of patients with clavicular fracture | At time of delivery
Number of patients with humeral fracture | At time of delivery
Number of patients with brachial plexus palsy | At time of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Chasen, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Prebyterian Hospital Weill Cornell, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No